CLINICAL TRIAL: NCT04688658
Title: A Phase I/II Study of PI3Kγδ Inhibitor Duvelisib in Combination With Nivolumab in Patients With Advanced Unresectable Melanoma Who Have Progressed on Anti-PD1 Therapy
Brief Title: Duvelisib in Combination With Nivolumab in Patients With Advanced Unresectable Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Secura Bio, Inc. discontinued support of the trial.
Sponsor: John Kirkwood (Other)
Collaborators: Secura Bio, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, John Kirkwood, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-155
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Unresectable Melanoma
Keywords: Anti-PD-1 monoclonal antibody (mAb)
MeSH Terms: interventions — Nivolumab; Axitinib; duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Duvelisib plus Nivolumab (Experimental): Phase 1: Duvelisib will be taken orally in doses from 15mg once a day, 25mg once a day or 25mg twice a day, 12 hours a part, to determine the recommended dose for the Phase II study when combined with nivolumab.
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks if deemed appropriate by the study doctor.
  Phase II: The Recommended Phase II dosage of duvelisib administered will not be determined until Phase I is completed.
  Nivolumab, 480mg, IV, every 4 weeks, for up to 1 year.
  Interventions: Drug: Nivolumab; Drug: Duvelisib

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Other Names: Opdivo; AG013736
Drug: Duvelisib — Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
  Other Names: Copiktra

SUMMARY:
This trial is a Phase I/II study in which a combination of duvelisib and nivolumab will be used to treat a total of patients diagnosed with advanced unresectable melanoma who have progressed on anti-PD1 therapy. The Recommended Phase II Dose of oral duvelisib will be determined and administered with intravenous nivolumab 480mg for up to 1 year or until the patient's disease does not progress or the patient experiences unacceptable side effects to treatment.

DETAILED DESCRIPTION:
This trial will study of PI3Kγδ inhibitor duvelisib in combination with nivolumab in patients with advanced unresectable melanoma who have progressed on anti-PD1 therapy. In the Phase I part of the study (18) patients will be administered nivolumab 480mg intravenously and duvelisib orally in doses from 15mg once a day to 25mg twice a day to determine the recommended dose for the Phase II part of the study. In the Phase II study patients will be administered nivolumab 480mg intravenously and duvelisib orally (dose not determined until the Phase 1 study is completed) up to 1 year as long as their disease doesn't progress or have unacceptable side effects to the study drugs. This trial will attempt to determine whether duvelisib acts as an immunomodulator, to shift the TME from an immunosuppressive to an immunostimulatory setting, to overcome acquired resistance in anti-PD1 treated patients. The phase I portion of the study is uniquely designed to find the ideal dose of duvelisib as an immunomodulator, which is suspected to be lower than the previously determined maximum tolerated dose (MTD) of duvelisib in lymphoma studies.

ELIGIBILITY:
Inclusion Criteria:

* AJCC 8th edition criteria for unresectable stage IIIB, stage IIIC, stage IIID or stage IV melanoma who have received at least 3 months of prior treatment with an anti-PD1 or anti-PDL1 antibody and who have progressed on this treatment. Patients who have received a combination anti-PD1 and anti-CTLA4 therapy who exhibit progression at this interval are also permitted. There are no restrictions regarding time since last anti-PD1 treatment, or number of therapies after anti-PD1.
* Age ≥ 18 years
* ECOG performance status ≤ 2 or Karnofsky ≥ 60%
* Patients must have normal organ and bone marrow function as defined below:

  * Hemoglobin ≥9.0 g/dL
  * Absolute neutrophil count ≥1500 cells/µL
  * Platelets ≥100,000 cells/µL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). Patients with Gilbert's syndrome must have normal direct bilirubin
  * AST/ALT ≤2.5x ULN in subjects with liver metastasis, must be within normal limits for those without liver metastasis
  * Creatinine < 1.5 mg/dL
* For patients with actionable BRAF mutations, treatment with BRAF and MEK inhibitors prior to initiation on trial is recommended, unless patients are intolerant of therapy or choose not to pursue BRAF targeted therapy.
* Patients must have measurable disease, defined as at least one tumor lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥10mm with CT scan, MRI or by calipers if documented on clinical exam. If patients have a single lesion, the lesion must be amenable to biopsy without interfering with radiographic assessment as determined by one of the co-PIs.
* Duvelisib and nivolumab therapy may be harmful for a developing fetus. Women of child bearing potential (WCBP) must have a negative urine or serum β human chorionic gonadotropin (βhCG) pregnancy test within 7 days before starting treatment. WCBP and men must agree to use highly effective contraception (pharmacologic birth control, barrier methods or abstinence) prior to study entry and for the duration of study participation through 5 months after the last dose of study medication. Should a woman become pregnant while she or her partner are participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use highly effective contraception prior to the study, for the duration of study participation and 12 weeks following the last dose.
* WCBP defined as a sexually mature woman who as not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months for women >55 years of age
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients with known or suspected CNS metastases with are excluded, unless the following criteria are met:

  * Subjects have controlled brain metastasis, defined as metastases without radiographic progression for at least 4 weeks following treatment with stereotactic radiation and/or surgical treatment at the time of randomization
  * Subjects must be off steroids without symptoms of CNS disease for at least 2 weeks prior to treatment
  * Subjects with signs or symptoms of brain metastasis are not eligible unless brain metastasis is ruled out by computed tomography or magnetic resonance imaging
* Patients with uveal or mucosal melanoma are excluded
* Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders such as vitiligo, alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with history of chronic liver disease, veno-occlusive disease, active alcohol abuse or illicit drug use other than marijuana or its derivatives
* Uncontrolled or significant cardiovascular disease including but not limited to the following:

  * Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
  * Uncontrolled angina within the 3 months prior to consent
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes, or poorly controlled atrial fibrillation)
  * History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled deep venous thrombosis, etc)
  * Cardiovascular disease-related requirement for daily supplemental oxygen
  * Subjects with history of myocarditis, regardless of etiology
  * Baseline left ventricular ejection fraction (LVEF) <45%. ECHO/MUGA not required at screening unless history of significant cardiac history.
  * QTc prolongation > 500 msec
* Uncontrolled or significant pulmonary disease including but not limited to the following:

  * Obstructive or restrictive lung disease requiring home oxygen
  * Hospitalization with chronic obstructive pulmonary disease (COPD) exacerbation within the last 6 months
  * History or concurrent condition of interstitial lung disease of any severity
  * Prior history of pneumonitis of grade II or higher, regardless of cause
  * Patients with diagnosis of obstructive sleep apnea (OSA) who are compliant with prescribed therapy (nocturnal O2, CPAP or BiPAP) are allowed on study
* Uncontrolled or significant infectious disease including but not limited to the following:

  * Ongoing treatment for systemic bacterial, fungal or viral infection at screening
  * Subjects are not excluded for antimicrobial, antifungal or antiviral prophylaxis if other inclusion/exclusion criteria are met
  * Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection (i.e., subjects with known history of detectable viral load)
  * Infection with hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or human T-lymphotropic virus type 1
  * Subjects with a positive hepatitis B surface antigen [HBsAg] or hepatitis C antibody [HCV Ab] will be excluded, unless documented treatment and resolution of hepatitis C treatment Subjects with a positive hepatitis B core antibody (HBcAb) must have negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) assay to be eligible, must receive prophylaxis with entecavir (or equivalent) concomitant with duvelisib treatment, and must be periodically monitored for HBV reactivation by institutional guidelines. If unable to receive prophylaxis, then case will be discussed with investigators to determine eligibility.
  * History of tuberculosis treatment within 2 years prior to enrollment
* Patients with history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
* Ongoing chronic treatment with immunosuppressants (e.g. cyclosporine) or systemic steroids > 10mg of prednisone or equivalent once daily. Topical and inhaled steroids are allowed.
* Subjects with other uncontrolled medical conditions or other illnesses, laboratory findings or other factors that would, in the investigator's judgment, increase the risk to the subject associated with his or her participation in the study.
* Patients who are receiving other investigational therapies will be excluded
* Patients who had a history of life-threatening toxicity related to prior immune therapy (e.g. anti-CTLA-4, anti-PD1 or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are well controlled an unlikely to be an issue with standard countermeasures (e.g. endocrine disorders managed by hormone replacement).
* Subjects with a history of grade II or greater immune-mediated colitis. Patients whose toxicity was clearly attributable to anti-CTLA-4 treatment (tolerated anti-PD1 after receiving anti-CTLA4) may still be allowed on trial.
* Subjects with a history of grade II or greater pneumonitis or transaminitis.
* Prior treatments with PI3K inhibitors
* Subject has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone therapy with curative intent, or treated in situ cervical cancer for which there is appropriate ongoing surveillance
* Subject had therapy with radiation, surgery or chemotherapy within 4 weeks prior to time of consent and/or has not recovered from adverse events to due to prior therapy. Subjects should be adequately recovered from all toxicities, complications, or acute illnesses prior to starting investigational therapy.
* A maximum of three patients who have received talimogene laherparepvec (T-vec) as prior therapy will be allowed to enroll in the Phase II portion of the study. However, study-related biopsies must be performed at a disease site that was not injected with T-vec or adjacent to a T-vec injection site.
* Subjects who are unable or unwilling to take prophylaxis for Pneumocystis jirovecii, human simplex virus (HSV) or herpes zoster (VZV) at time of screening
* Subjects with known hypersensitivity to duvelisib and/or its excipients: Microcrystalline cellulose and magnesium stearate
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
* Subjects who are unable or unwilling to comply with restrictions and prohibited activities and treatments
* Subjects who are unable or unwilling to undergo venipuncture or tolerate venous access
* Subjects with prior surgery and/or chronic gastrointestinal dysfunction that may affect drug absorption, such as gastric bypass, gastrectomy, malabsorption, inflammatory bowel disease, chronic diarrhea
* Concurrent administration of medications or foods that are strong inhibitors of inducers of cytochrome p450 3A (CYP3A) within 2 weeks prior to study intervention. Duvelisib can increase exposure to CYP3A4 substrates; consider dose reduction of such substrates and monitor for signs of toxicities of co-administered sensitive CYP3A substrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkwood, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Phase 1: 25 mg BID Duvelisib and Phase II arms.
Groups:
- Duvelisib (15mg) + Nivolumab (240mg): Phase 1:
  Duvelisib,15mg once a day, 12 hours a part, to determine the recommended dose for the Phase II study when combined with nivolumab.
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor)
  Phase II: The Recommended Phase II dosage of duvelisib administered will not be determined until Phase I is completed.
  Nivolumab, 480mg, IV, every 4 weeks, for up to 1 year.
  Nivolumab: Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Duvelisib: Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
- Duvelisib (25mg) + Nivolumab (240mg): Phase 1:
  Duvelisib,25mg once a day, 12 hours a part, to determine the recommended dose for the Phase II study when combined with nivolumab.
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor)
Period: Overall Study
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg) | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Median (Full Range); unit: years] | 66.00 [51.00 to 79.00] | 65.50 [49.00 to 77.00] | 66.00 [49.00 to 79.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
BRAF Status [Count of Participants; unit: Participants] — BRAF mutations are found in roughly half of melanomas. Medications that target these mutations have improved survival rates of metastatic melanoma setting.
  Participants
    Mutant | 2 | 0 | 2
    Wild Type (WT) | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: DLTs by Phase I Dose of Duvelisib With Nivolumab
Description: Number of patients experiencing acute dose limiting toxicities (DLTs) and laboratory abnormalities considered possibly related to study treatment, occurring from the initial dose of duvelisib + nivolumab through day 28 of treatment (acute) or toxicities occurring from day 29 through 28 days after completion of treatment (late toxicities). DLTs are defined using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 56 days (per patient)
Population: Treated patients evaluated for dose limiting toxicities.
Measure: Number; unit: participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

2. Primary Outcome: Best Overall Response
Description: Best Response per RECIST v1.1: Completed Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis); Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum diameters while on study. Progressive Disease (PD): ≥20% (relative) increase in sum of diameters of target lesions referencing smallest sum on study (includes baseline sum if is smallest on study) and, the sum must also demonstrate an absolute increase of at least 5 mm; appearance of one or more new lesions.
Time Frame: Up to 29 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- Duvelisib (15mg) + Nivolumab (240mg): Duvelisib,15mg once a day, 12 hours a part
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor for up to 1 year)
  Nivolumab: Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Duvelisib: Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
- Duvelisib (25mg) + Nivolumab (240mg): Duvelisib, 25mg once a day, 12 hours a part
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor for up to 1 year)
  Nivolumab: Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Duvelisib: Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
Participants
  Partial Response (PR) | 1 | 0
  Stable Disease (SD) | 1 | 1
  Progressive Disease (PD) | 3 | 3

3. Primary Outcome: Best Overall Response Rate (ORR)
Description: Proportion of patients with a Best Response (CR+PR)/(CR+PR+SD+PD) per RECIST v1.1 of Completed Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis); or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 29 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
proportion of patients | 0.20 [0.0051 to 0.7164] | 0.0 [0 to 0.6024]

4. Primary Outcome: Change in CD 8+ TIL Frequency
Description: CyTek flow cytometry will be used to evaluate tumor-infiltrating cells in PBMCs and tumor tissue for the increased frequency (proliferation) and activation of CD8+ TILs. Proliferation of CD8+ TIL cells correlate with improved survival in patients with melanoma.
Time Frame: Baseline to Week 4
Population: Treated patients who provided samples for CD 8+ TIL testing.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of cells
  Total CD8 T-cells (%CD45) | -0.87 (2.91) | 2.66 (3.65)
  Total Cycling CD8 (%Ki67+) | 2.86 (1.94) | 10.26 (23.11)
  NAV. %CD8 | -2.52 (6.07) | -1.44 (6.61)
  TCM. %CD8 | 0.84 (3.89) | -0.22 (5.13)
  TEM %CD8 | 2.92 (4.60) | 1.46 (4.98)
  TEMRA. %CD8 | -1.25 (1.94) | -0.88 (7.09)

5. Secondary Outcome: Clinical Benefit
Description: Complete response [CR], partial response [PR] or stable disease [SD], per RECIST v1.1 criteria . Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis);PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): ≥20% (relative) increase in sum of diameters of target lesions referencing smallest sum on study (includes baseline sum if is smallest on study) and, the sum must also demonstrate an absolute increase of at least 5 mm; appearance of one or more new lesions.
Time Frame: At Week 12
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
Participants
  Partial Response (Week 12) | 1 | 0
  Stable Disease (Week 12) | 0 | 1
  Progressive Disease (Week 12) | 4 | 3

6. Secondary Outcome: Clinical Benefit
Description: Complete response [CR], partial response [PR], stable disease [SD], per RECIST v1.1 criteria . Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis);PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): ≥20% (relative) increase in sum of diameters of target lesions referencing smallest sum on study (includes baseline sum if is smallest on study) and, the sum must also demonstrate an absolute increase of at least 5 mm; appearance of one or more new lesions.
Time Frame: At Week 24
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
Participants | 1 | 0

7. Secondary Outcome: Clinical Benefit
Description: as for outcome 6
Time Frame: At Week 48
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
Participants | 1 | 0

8. Secondary Outcome: Clinical Benefit Rate
Description: Proportion of patients (CR + PR + SD)/(CR + PR + SD +PD) Complete response [CR], partial response [PR], stable disease [SD], per RECIST v1.1 criteria. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis);PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): ≥20% (relative) increase in sum of diameters of target lesions referencing smallest sum on study (includes baseline sum if is smallest on study) and, the sum must also demonstrate an absolute increase of at le
Time Frame: At Week 12
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
proportion of patients | 0.20 [0.0051 to 0.7164] | 0.25 [0.0063 to 0.8059]

9. Secondary Outcome: Acute Adverse Events at Least Possibly Related to Treatment
Description: Number and percentage of Acute adverse events as graded by CTCAE v5.0 in patients at each dosing interval and in the expansion cohort. Toxicity events include those that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Time Frame: Up to 4 weeks
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 7 | 6
Participants
  Anemia | 1 | 0
  Diarrhea | 1 | 0
  Vomiting | 0 | 1
  Chills | 0 | 1
  Fever | 0 | 1
  CD4 lymphocytes decreased | 0 | 1
  Hyponatremia | 1 | 0
  Myalgia | 1 | 0

10. Secondary Outcome: Late Adverse Events at Least Possibly Related to Treatment
Description: Number and percentage of Late occurring adverse events as graded by CTCAE v5.0 in patients at each dosing interval and in the expansion cohort. Toxicity events include those that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Time Frame: Beginning at 4 weeks after start of treatment, up to 14 months
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 7 | 6
Participants
  Hyperthyroidism | 2 | 0
  Diarrhea | 0 | 1
  Vomiting | 0 | 1
  Hypothyroidism | 0 | 1
  Dry mouth | 0 | 1
  CD4 lymphocytes decreased | 1 | 0
  Fatigue | 2 | 0
  Hepatic failure | 0 | 1
  Alanine aminotransferase increased | 3 | 3
  Alkaline phosphatase increased | 1 | 1
  Aspartate aminotransferase increased | 3 | 3
  Blood bilirubin increased | 0 | 1
  Lymphocyte count decreased | 0 | 1
  Neutrophil count decreased | 0 | 1
  White blood cell decreased | 0 | 1
  Anorexia | 1 | 0
  Generalized muscle weakness | 0 | 1
  Proteinuria | 1 | 0
  Hypertension | 1 | 0

11. Secondary Outcome: Treatment Related Adverse Events
Description: Number of patients who experienced adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Time Frame: Up to 42.5 months
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 7 | 6
Participants | 5 | 5

12. Secondary Outcome: Treatment Related Serious Adverse Events
Description: Number of patients who experienced serious adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Time Frame: Up to 42.5 months
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 7 | 6
Participants | 3 | 1

13. Secondary Outcome: Treatment-related Grade 3 or Higher AE
Description: Number of Patients with Treatment-related Grade 3 or Higher AE per CTCAE v5.0
Time Frame: Up to 42.5 months
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 7 | 6
Participants | 4 | 4

14. Secondary Outcome: Number of Patients With Clinical Response
Description: Number of patients with Complete Response (CR) or Partial Response (PR) until the first time at which progressive disease is objectively documented per RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumormarker level. All lymph nodes must be non-pathological in size (<10mm short axis);PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 36 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number; unit: participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 4
participants | 1 | 0

15. Secondary Outcome: Overall Survival (OS)
Description: The (median) length of time from the start of treatment that patients remain alive, until death from any cause. Patients who are alive will be censored at the time of the last follow-up.
Time Frame: Up to 25 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
  Among the 13 enrolled patients, 3 (2 in the 15 mg arm and 1 in the 25mg arm) were not evaluable as, per protocol, no duvelisib pills were returned for these patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
months | 13.5 [12.2 to NA] — Upper bound of 95%CI not reached due small sample size and the rapidly decreasing number of patients at risk over time | 4.9 [3.9 to NA] — Upper bound of 95%CI not reached due small sample size and the rapidly decreasing number of patients at risk over time

16. Secondary Outcome: 6-month Overall Survival (OS)
Description: The percentage of patients alive at 6 months the start of treatment until death from any cause.
Time Frame: At 6 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Duvelisib (15mg) + Nivolumab (240mg): Duvelisib,15mg once a day, 12 hours a part
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor for up to one year)
  Nivolumab: Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Duvelisib: Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of patients | 80.0 [51.6 to 100.0] | 40.0 [13.7 to 100.0]

17. Secondary Outcome: 12-month Overall Survival (OS)
Description: The percentage of patients alive at 12 months the start of treatment until death from any cause.
Time Frame: At 12 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of patients | 80.0 [51.6 to 100.0] | 20.0 [3.5 to 100.0]

18. Secondary Outcome: 18-month Overall Survival (OS)
Description: The percentage of patients alive at 18 months the start of treatment until death from any cause.
Time Frame: At 18 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of patients | 40.0 [13.7 to 100.0] | NA [NA to NA] — All patients either experience event or were censored before this timepoint

19. Secondary Outcome: Overall Survival (OS) - Total Population
Description: as for outcome 15
Time Frame: Up to 25 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Duvelisib (15mg and 25mg) + Nivolumab (240mg): Duvelisib,15mg or 25mg once a day, 12 hours a part
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor for up to one year)
  Nivolumab: Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Duvelisib: Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
months | 9.9 [3.9 to NA] — Upper bound of 95% CI not reached due to limited number of events.

20. Secondary Outcome: 6-month Overall Survival (OS) - Total Population
Description: The percentage of patients alive at 6 months the start of treatment until death from any cause.
Time Frame: At 6 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
percentage of patients | 60.0 [36.2 to 99.5]

21. Secondary Outcome: 12-month Overall Survival (OS) - Total Population
Description: The percentage of patients alive at 12 months the start of treatment until death from any cause.
Time Frame: At 12 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
percentage of patients | 50.0 [26.9 to 92.9]

22. Secondary Outcome: 18-month Overall Survival (OS) -Total Population
Description: The percentage of patients alive at 18 months the start of treatment until death from any cause.
Time Frame: At 18 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
percentage of patients | 30.0 [11.6 to 77.3]

23. Secondary Outcome: Progression-free Survival (PFS)
Description: The (median) length of time from the initial date of treatment to the date of documented progression, or the date of death due to any cause (in the absence of progression, whichever occurs first), with progression defined by RECIST v1.1. PerRECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 36 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Duvelisib (15mg) + Nivolumab (240mg): Duvelisib, 15mg once a day, 12 hours a part
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor for up to 1 year)
  Nivolumab: Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Duvelisib: Duvelisib is a potent inhibitor of both γ and δ isoforms. Duvelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
months | 2.8 [2.8 to NA] — Upper bound of 95%CI not reached due to limited number of events | 3.0 [2.8 to NA] — Upper bound of 95%CI not reached due to limited number of events

24. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: The percentage of patients whose disease does not progress from initial date of treatment to at 6 months, with progression defined by RECIST v1.1. PerRECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: At 6 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of participants | 20 [3.5 to 100.00] | 0 [NA to NA] — At the 6-month timepoint, all patients on the 25mg dose experienced an event.

25. Secondary Outcome: 12-month Progression-free Survival (PFS)
Description: The percentage of patients whose disease does not progress from initial date of treatment to at 12 months, with progression defined by RECIST v1.1. PerRECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: At 12 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of participants | 0 [NA to NA] — At the 12-month timepoint, all patients on the experienced an event. | 0 [NA to NA] — At the 12-month timepoint, all patients on the experienced an event.

26. Secondary Outcome: 18-month Progression-free Survival (PFS)
Description: The percentage of patients whose disease does not progress from initial date of treatment to at 18 months, with progression defined by RECIST v1.1. PerRECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: At 18 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of participants | 0 [NA to NA] — At the 18-month timepoint, all patients experienced an event. | 0 [NA to NA] — At the 18-month timepoint, all patients experienced an event.

27. Secondary Outcome: Progression-free Survival (PFS) - Total Population
Description: as for outcome 23
Time Frame: Up to 36 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
months | 2.8 [2.6 to NA] — Upper bound of 95% CI not reached due to limited number of events.

28. Secondary Outcome: 6-month Progression-free Survival (PFS) - Total Population
Description: The percentage of patients whose disease does not progress from initial date of treatment to at 6 months, with progression defined by RECIST v1.1. Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: At 6 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
percentage of patients | 10.0 [1.6 to 64.2]

29. Secondary Outcome: 12-month Progression-free Survival (PFS) - Total Population
Description: as for outcome 25
Time Frame: At 12 months
Population: Patients who received at least one cycle of the treatment and at least one efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
percentage of patients | 0 [NA to NA] — At the 12-month timepoint, all patients from both dose levels had experienced progression or death before this timepoint; therefore, no patients remained progression-free at 12 months.

30. Secondary Outcome: 18-month Progression-free Survival (PFS) - Total Population
Description: as for outcome 26
Time Frame: At 18 months
Population: Treated patients who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib (15mg and 25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 10
percentage of participants | 0 [NA to NA] — At the 18-month timepoint, all patients from both dose levels had experienced progression or death before this timepoint; therefore, no patients remained progression-free at 18 months.

31. Other Pre Specified Outcome: Immune Cell Function
Description: Evaluation of peripheral blood mononuclear cells (PBMCs) using CyTek flow cytometry.
Time Frame: Baseline (prior to treatment), at 12 weeks after start of treatment; Up to 2 years (cohort)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Immune Cell Function
Description: Evaluation of tumor-infiltrating cells from using CyTek flow cytometry.
Time Frame: Baseline (prior to treatment), at 12 weeks after start of treatment; Up to 2 years (cohort)
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Tumor Microenvironment (TME)
Description: Changes in the immune cell population using Vectra imaging.
Time Frame: Baseline (prior to treatment), at 12 weeks after start of treatment; Up to 2 years (cohort)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Mechanism of Anti-PD1 Resistance
Description: Changes in gene expression in the tumor using Nanostring gene profiling.
Time Frame: Baseline (prior to treatment), at 12 weeks after start of treatment; Up to 2 years (cohort)
Reporting Status: Not Posted

35. Primary Outcome: Change in CD 8+ TIL Frequency
Description: as for outcome 4
Time Frame: Baseline to Week 12
Population: Treated patients who provided samples for CD 8+ TIL testing.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of cells
  Total CD8 T-cells (%CD45) | 4.05 (5.03) | -1.63 (3.58)
  Total Cycling CD8 (%Ki67+) | 15.86 (24.96) | 0.45 (3.70)
  NAV. %CD8 | -3.79 (4.80) | -1.68 (2.37)
  TCM. %CD8 | -0.15 (3.23) | -8.91 (3.41)
  TEM %CD8 | 7.97 (6.60) | 6.60 (6.65)
  TEMRA. %CD8 | -4.06 (8.10) | 4.00 (0.85)

36. Primary Outcome: Change in CD 8+ TIL Frequency
Description: as for outcome 4
Time Frame: Week 4 to Week 12
Population: Treated patients who provided samples for CD 8+ TIL testing.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
Number analyzed (Participants) | 5 | 5
percentage of cells
  Total CD8 T-cells (%CD45) | 4.11 (4.59) | -2.69 (0.69)
  Total Cycling CD8 (%Ki67+) | 12.52 (26.54) | 2.92 (8.39)
  NAV. %CD8 | 1.44 (2.19) | -1.70 (5.51)
  TCM. %CD8 | -1.88 (3.02) | -13.26 (6.73)
  TEM %CD8 | 4.03 (5.85) | 6.75 (6.86)
  TEMRA. %CD8 | -3.62 (6.62) | 8.20 (5.37)

ADVERSE EVENTS:
Time Frame: Adverse events data collected for up to 42.5 months for the study population.
Groups:
- Duvelisib (25mg) + Nivolumab (240mg): Phase 1:
  Duvelisib, 25mg once a day, 12 hours a part, to determine the recommended dose for the Phase II study when combined with nivolumab.
  Nivolumab, 240mg, IV, every 2 weeks for the first four cycles; thereafter it may be switched to 480mg, IV, once every 4 weeks (if deemed appropriate by the study doctor)
Arm/Group | Duvelisib (15mg) + Nivolumab (240mg) | Duvelisib (25mg) + Nivolumab (240mg)
All-Cause Mortality (participants affected / at risk) | 7/7 | 5/6
Serious Adverse Events (participants affected / at risk) | 6/7 | 4/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (15mg) + Nivolumab (240mg) (N=7) | Duvelisib (25mg) + Nivolumab (240mg) (N=6)
Atrial fibrillation (CARDIAC DISORDERS) | 1 | 0
Diarrhea (GASTROINTESTINAL DISORDERS) | 1 | 0
Retroperitoneal hemorrhage (GASTROINTESTINAL DISORDERS) | 1 | 0
Vomiting (GASTROINTESTINAL DISORDERS) | 1 | 0
Death NOS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 | 0
Hepatic failure (HEPATOBILIARY DISORDERS) | 1 | 0
Covid (INFECTIONS AND INFESTATIONS) | 1 | 0
Lung infection (INFECTIONS AND INFESTATIONS) | 0 | 1
Sepsis (INFECTIONS AND INFESTATIONS) | 0 | 1
Alanine aminotransferase increased (INVESTIGATIONS) | 2 | 1
Aspartate aminotransferase increased (INVESTIGATIONS) | 2 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) -Other, specifyBrain |Neoplasm (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 | 1
Edema cerebral (NERVOUS SYSTEM DISORDERS) | 0 | 1
Encephalopathy (NERVOUS SYSTEM DISORDERS) | 0 | 1
Lethargy (NERVOUS SYSTEM DISORDERS) | 0 | 1
Seizure (NERVOUS SYSTEM DISORDERS) | 0 | 1
Confusion (PSYCHIATRIC DISORDERS) | 0 | 2
Acute kidney injury (RENAL AND URINARY DISORDERS) | 1 | 0
Respiratory failure (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 0
sternectomy with reconstruction (SURGICAL AND MEDICAL PROCEDURES) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (15mg) + Nivolumab (240mg) (N=7) | Duvelisib (25mg) + Nivolumab (240mg) (N=6)
Anemia (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 4 | 5
Eosinophilia (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 | 1
Leukocytosis (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 | 1
Pericardial effusion (CARDIAC DISORDERS) | 1 | 0
Sinus bradycardia (CARDIAC DISORDERS) | 1 | 0
Sinus tachycardia (CARDIAC DISORDERS) | 3 | 1
Hyperthyroidism (ENDOCRINE DISORDERS) | 1 | 2
Dry eye (EYE DISORDERS) | 1 | 0
Abdominal pain (GASTROINTESTINAL DISORDERS) | 1 | 0
Constipation (GASTROINTESTINAL DISORDERS) | 4 | 1
Diarrhea (GASTROINTESTINAL DISORDERS) | 1 | 0
Dry mouth (GASTROINTESTINAL DISORDERS) | 1 | 0
Nausea (GASTROINTESTINAL DISORDERS) | 2 | 3
Vomiting (GASTROINTESTINAL DISORDERS) | 0 | 3
Chills (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1
Edema limbs (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 1
Fatigue (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4 | 3
Fever (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 1
Pain (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 | 1
Fall (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 3
lymph node pain (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1
restlessness (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1
Back Pain (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 2
Upper respiratory infection (INFECTIONS AND INFESTATIONS) | 0 | 1
Bruising (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 1
Pain - Surgical (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 0
Tumor |Pain - |Chest (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 0
Generalized edema (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 0
Non-cardiac chest pain (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 0
Pneumonia (INFECTIONS AND INFESTATIONS) | 1 | 0
Sepsis (INFECTIONS AND INFESTATIONS) | 1 | 0
Thrush (INFECTIONS AND INFESTATIONS) | 1 | 1
Urinary tract infection (INFECTIONS AND INFESTATIONS) | 1 | 1
Activated partial thromboplastin time prolonged (INVESTIGATIONS) | 1 | 1
Alanine aminotransferase increased (INVESTIGATIONS) | 1 | 2
Alkaline phosphatase increased (INVESTIGATIONS) | 2 | 2
Aspartate aminotransferase increased (INVESTIGATIONS) | 2 | 2
Blood bilirubin increased (INVESTIGATIONS) | 1 | 1
Blood lactate dehydrogenase increased (INVESTIGATIONS) | 4 | 3
Cardiac troponin I increased (INVESTIGATIONS) | 2 | 0
CD4 lymphocytes decreased (INVESTIGATIONS) | 0 | 2
Creatinine increased (INVESTIGATIONS) | 3 | 2
INR increased (INVESTIGATIONS) | 1 | 0
Elevated CRP (INVESTIGATIONS) | 0 | 1
Partial thromboplastin time increased (INVESTIGATIONS) | 0 | 1
Prothrombin time increased (INVESTIGATIONS) | 0 | 1
Lymphocyte count decreased (INVESTIGATIONS) | 5 | 2
Neutrophil count decreased (INVESTIGATIONS) | 1 | 1
Platelet count decreased (INVESTIGATIONS) | 1 | 0
Weight gain (INVESTIGATIONS) | 1 | 0
White blood cell decreased (INVESTIGATIONS) | 2 | 1
Anorexia (METABOLISM AND NUTRITION DISORDERS) | 3 | 4
Dehydration (METABOLISM AND NUTRITION DISORDERS) | 2 | 1
Hypercalcemia (METABOLISM AND NUTRITION DISORDERS) | 2 | 0
Hyperglycemia (METABOLISM AND NUTRITION DISORDERS) | 2 | 5
Hyperkalemia (METABOLISM AND NUTRITION DISORDERS) | 3 | 1
Hypermagnesemia (METABOLISM AND NUTRITION DISORDERS) | 1 | 0
Hypernatremia (METABOLISM AND NUTRITION DISORDERS) | 1 | 0
Hypertriglyceridemia (METABOLISM AND NUTRITION DISORDERS) | 1 | 0
Hypoalbuminemia (METABOLISM AND NUTRITION DISORDERS) | 3 | 4
Hypocalcemia (METABOLISM AND NUTRITION DISORDERS) | 2 | 3
Hypoglycemia (METABOLISM AND NUTRITION DISORDERS) | 1 | 0
Hypokalemia (METABOLISM AND NUTRITION DISORDERS) | 2 | 3
Hypomagnesemia (METABOLISM AND NUTRITION DISORDERS) | 2 | 2
Hyponatremia (METABOLISM AND NUTRITION DISORDERS) | 6 | 6
Hypophosphatemia (METABOLISM AND NUTRITION DISORDERS) | 2 | 1
Back pain (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 | 0
Generalized muscle weakness (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 | 1
Myalgia (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 | 0
Dysphasia (NERVOUS SYSTEM DISORDERS) | 1 | 0
Lethargy (NERVOUS SYSTEM DISORDERS) | 2 | 0
Somnolence (NERVOUS SYSTEM DISORDERS) | 1 | 0
Agitation (PSYCHIATRIC DISORDERS) | 2 | 0
Dizziness (NERVOUS SYSTEM DISORDERS) | 0 | 1
Dysgeusia (NERVOUS SYSTEM DISORDERS) | 0 | 1
Headache (NERVOUS SYSTEM DISORDERS) | 0 | 2
Agitation (NERVOUS SYSTEM DISORDERS) | 0 | 1
Anxiety (PSYCHIATRIC DISORDERS) | 2 | 1
Confusion (PSYCHIATRIC DISORDERS) | 1 | 0
Delirium (PSYCHIATRIC DISORDERS) | 0 | 1
Acute kidney injury (RENAL AND URINARY DISORDERS) | 0 | 1
Chronic kidney disease (RENAL AND URINARY DISORDERS) | 0 | 1
Hematuria (RENAL AND URINARY DISORDERS) | 0 | 2
Proteinuria (RENAL AND URINARY DISORDERS) | 0 | 2
Glucosuria (RENAL AND URINARY DISORDERS) | 1 | 0
Hematuria (RENAL AND URINARY DISORDERS) | 1 | 0
Proteinuria (RENAL AND URINARY DISORDERS) | 3 | 0
Urine discoloration (RENAL AND URINARY DISORDERS) | 1 | 0
Reproductive system and breast disorders - |Other, specifyLabial |Lesion |Pain (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 | 0
Reproductive system and breast disorders - |Other, specifypain (labia) (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 | 0
Cough (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 1
Epistaxis (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 0
Dyspnea (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1
Respiratory, thoracic and mediastinal disorders - |Other, specifyHemoptysis (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1
Rash maculo-papular (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 1
Surgical and medical procedures - |Other, specifyCraniotomy (SURGICAL AND MEDICAL PROCEDURES) | 0 | 1
Rash acneiform (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 | 0
deep tissue pressure injury on buttocks (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 | 0
Hematoma (VASCULAR DISORDERS) | 1 | 0
Hypertension (VASCULAR DISORDERS) | 3 | 3
Hypotension (VASCULAR DISORDERS) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04688658/Prot_SAP_000.pdf